CLINICAL TRIAL: NCT03511703
Title: A Randomized Clinical Study of The Treatment of Postoperative Adjuvant Apatinib vs. TACE in Hepatocellular Carcinoma Patients
Brief Title: The Study of The Treatment of Postoperative Adjuvant Apatinib vs. TACE in Hepatocellular Carcinoma Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, TaoBai, Researcher, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GuangxiMU-HCCop
Record Dates: First submitted 2018-04-18; First posted 2018-04-30 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — apatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib (Experimental)
  Interventions: Drug: Apatinib
- TACE (Other)
  Interventions: Drug: Chemotherapy drugs+Iodized oil

INTERVENTIONS:
Drug: Apatinib — Apatinib, a small molecule anti-angiogenic targeted drug that has been demonstrated to be safe and effective after failure of standard chemotherapy for advanced gastric cancer, has been initially successful in phase II clinical trials for the treatment of unresectable advanced HCC patients. The efficacy of ralfiny in the treatment of Oriental population (ORIENTAL study) is better. The randomized, doubleblind, multi-center phase III clinical study of apatinib second-line treatment of advanced hepatocellular carcinoma showed a good efficacy and safety. Currently, Phase III clinical studies of apatinib in HCC patients undergoing systemic chemotherapy or sorafenib treatment have progressed. Initial results lso showed good efficacy and safety.
  Arms: Apatinib
Drug: Chemotherapy drugs+Iodized oil — Intra-arterial infusion chemotherapy for tumors, commonly used chemotherapy drugs include anthracyclines, platinum, etc.; chemotherapeutic drugs and embolic agents are mixed together and injected through the blood supply artery of the tumor. The most commonly used embolic agent for TACE treatment is a lipiodol emulsion. First infusion of some chemotherapy drugs, the general infusion time should not be <20 min. Then another part of the chemotherapeutic drugs and lipiodol were mixed into emulsions for embolization. The amount of lipiodol is generally 5-20 ml, not more than 30 ml.
  Arms: TACE

SUMMARY:
This study uses to suppress the growth of tumors, extend the patient's survival time and improve the quality of life as much as possible. Through the treatment, the patient is given the chance to undergo surgical resection, thereby more effectively prolonging the OS. Apatinib is a small-molecule VEGFR tyrosine kinase inhibitor. It mainly treats malignant tumors by inhibiting VEGFR and exerting anti-angiogenic effects. Preclinical studies have shown that its antitumor effect is better than that of the similar drug PTK787. Phase II studies of hepatocellular carcinoma have initially demonstrated the effectiveness and safety of apatinib in the treatment of advanced HCC. TACE embolized tumor artery blood supply to inhibit tumor growth and shrink tumors. Based on the therapeutic potential of apatinib, and TACE in their respective tumors, we designed a prospective exploratory clinical study of this patient with advanced liver cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years old;
2. HCC diagnosed by histopathology or cytology (including pathological margin positive lesions, residual positive lesions after DSA angiography, combined vascular tumor thrombus and/or biliary tumor thrombus, pathologically confirmed lymph node metastasis, and liver The tumor ruptured, adjacent organs were invaded, the number of tumors was ≥ 3, AFP did not fall to normal range at 2 months after operation, and pathologically confirmed vegf + or patients with microvascular invasion.
3. Child-Pugh Liver Function Rating: Grade A or better Grade B (≤ 7 points);
4. ECOG PS score: 0-1 points;
5. Expected survival period ≥ 12 weeks;
6. The normal function of the major organs is the following:

(1) Blood tests: HB≥90 g/L; ANC≥1.5×109/L; PLT≥60×109/L; (2) Biochemical tests: ALB ≥29 g/L; ALT and AST<2.5ULN; TBIL ≤ 2ULN; Creatinine ≤1.5ULN; (Child-Pugh can only have 2 points for both albumin and bilirubin) 7. Women of childbearing age must undergo a pregnancy test within 7 days prior to enrollment; 8. Subjects voluntarily joined the study, signed informed consent, and adhered well to follow-up.

Exclusion Criteria:

1. Have received systematic treatment in the past;
2. Hepatobiliary cell carcinoma and mixed cell carcinoma and fibrous lamellar cell carcinoma are known; in the past (within 5 years) or with other untreated malignant tumors, except for cured skin basal cell carcinoma and cervical carcinoma in situ;
3. Patients who are preparing for liver transplantation (except those who have previously undergone liver transplantation);
4. Ascites with clinical symptoms, which require therapeutic paracentesis or drainage;
5. People with high blood pressure who are unable to fall within the normal range after treatment with antihypertensive drugs (systolic blood pressure>140 mmHg, diastolic blood pressure>90 mmHg);
6. Arrhythmia with grade II or higher myocardial ischemia or myocardial infarction and poor control (including QMS interval men ≥450 ms, women ≥470 ms);
7. In accordance with NYHA criteria III-IV heart failure or cardiac ultrasound examination: LVEF (left ventricular ejection fraction) <50%;
8. Has a variety of factors that affect oral medications (such as inability to swallow, chronic diarrhea, and intestinal obstruction, which significantly affect drug intake and absorption);
9. In the past 6 months, there was a history of digestive tract bleeding or a clear tendency to gastrointestinal bleeding. For example, esophageal varices, local active ulcer lesions, fecal occult blood ≥ (++) may not enter the group. If fecal occult blood (+) requires gastroscopy;
10. Abdominal fistula, gastrointestinal perforation or abdominal abscess occurred within 28 days before participating in this study;
11. Coagulation abnormalities (INR> 1.5 or prothrombin time (PT)> ULN + 4 seconds) with a tendency to hemorrhage or receiving thrombolytic or anticoagulant therapy;
12. Patients with central nervous system metastases or known brain metastases have occurred;
13. Patients with objective evidence of previous and current history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, and severe impaired lung function;
14. Urine routine showed urinary protein ≥ ++ or confirmed 24-hour urinary protein quantification> 1.0 g;
15. Was treated with potent CYP3A4 inhibitors within 7 days before participating in the study or was treated with potent CYP3A4 inducer within 12 days prior to study participation;
16. Pregnancy or breastfeeding women; those with fertility who are unwilling or unable to take effective contraceptive measures;
17. There is a history of mental illness or abuse of psychotropic substances;
18. Patients with bone metastases who have received palliative radiotherapy (radiotherapy area> 5% bone marrow area) within 4 weeks before participating in the study;
19. Joint HIV-infected patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 years